CLINICAL TRIAL: NCT05418972
Title: A Phase 2, Open Label, Single Arm, Clinical Trial of Neoadjuvant Relatlimab and Nivolumab in High Risk, Clinical Stage II Cutaneous Melanoma
Brief Title: A Phase 2 Clinical Trial of Neoadjuvant Relatlimab and Nivolumab in High Risk, Clinical Stage II Cutaneous Melanoma
Acronym: Neo ReNi II
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma Institute Australia (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIA2022/CT/432, CA224-137
Record Dates: First submitted 2022-06-09; First posted 2022-06-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Stage II Melanoma
Keywords: Neoadjuvant; Nivolumab; Relatlimab; Pathological response; Biomarkers; Feasibility; Sentinel node biopsy; Lymphoscintigraphy; Single-photon emission computed tomography (SPECT)
MeSH Terms: conditions — Melanoma | interventions — relatlimab; Nivolumab; Opdualag

STUDY DESIGN:
Intervention Model Description: Open label, single arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant immunotherapy +/- Adjuvant immunotherapy (Experimental): NEOADJUVANT: All participants will receive neoadjuvant therapy with the fixed dose combination of intravenous relatlimab 160 mg and nivolumab 480 mg x 2 doses on days 1 and 29.
  SURGERY: All participants will have sentinel lymph node mapping and biopsy prior to a wide local excision of the primary melanoma between days 43 and 56.
  ADJUVANT: Participants with no pathological response or partial pathological response will receive the fixed dose combination of intravenous relatlimab 160 mg and nivolumab 480 mg for a further 11 doses.
  Interventions: Drug: Relatlimab and nivolumab fixed dose combination (FDC)

INTERVENTIONS:
Drug: Relatlimab and nivolumab fixed dose combination (FDC) — Lymphocyte activation gene-3 (LAG-3) and programmed death-1 (PD-1) are two distinct inhibitory immune checkpoints that are often co-expressed on tumor-infiltrating lymphocytes, thus contributing to tumor-mediated T-cell exhaustion. The combination of nivolumab (anti-PD-1) and relatlimab (anti-LAG-3) results in increased T-cell activation compared to the activity of either antibody alone.
  Other Names: Opdualag

SUMMARY:
Neoadjuvant therapy is feasible in stage II melanoma, and the dual inhibition of the distinct LAG-3 and PD-1 checkpoint pathways with relatlimab and nivolumab has a synergistic effect in the tumour microenvironment leading to a pathological response after 2 doses of therapy.

DETAILED DESCRIPTION:
The incidence of stage II melanoma is significantly higher than for later stages of the disease, but stage II patients account for approximately 50% of all those who subsequently develop metastatic disease and die. Stage II melanomas have a Breslow thickness greater than 1.0 mm, with no clinical evidence of nodal, satellite or distant metastases. Pathological staging requires evaluation of the regional node basin after lymphatic mapping and sentinel node biopsy (SNB), which is required for N categorization of all >T1 melanomas. Compared to stage III disease, stage IIB and IIC have a worse prognosis than stage IIIA melanomas. Stage IIC even share the same poor prognosis as stage IIIB.

Global management guidelines highlight the importance of an initial diagnostic biopsy to confirm the diagnosis of melanoma and to pathologically stage the tumour. After the diagnosis and Breslow thickness and other features have been established by histological assessment of the initial excision biopsy, the definitive management of primary cutaneous melanoma consists of surgical excision with a safety margin of surrounding skin and subcutaneous tissue. Sentinel lymph node biopsy (SNB) should be considered for melanomas ≥ 1 mm thickness (≥ 0.8 mm if ulcerated or other high-risk features) in which case lymphoscintigraphy must be performed just prior to wider excision of the primary melanoma site.

Despite the equivalent risk, the current standard of care for stage IIB/C melanoma is observation only although this is expected to change given the results from recent studies investigating adjuvant drug therapy in this stage. Importantly, systemic adjuvant therapy is standard for stage IIIB/C/D disease. Although patients with stage II disease contribute the largest population to melanoma-specific mortality, under the current treatment guidelines, these patients represent a population less likely to be treated in the adjuvant setting and have no representation in the neoadjuvant setting.

Patients at low risk of recurrence with stage IIA disease (tumour >2-4 mm in thickness without ulceration [T3a], or >1 to 2 mm in thickness with ulceration [T2b]), have a high probability to be cured by surgery alone. However, the 5-year melanoma-specific survival (MSS) in stage IIA is 94%, which is comparable to the 93% of stage IIIB; patients with stage IIIA disease have a better prognosis than those with stage IIC disease. Patients diagnosed with higher risk stage IIB/C disease have thicker melanomas > 2.0 mm with ulceration, and > 4.0 mm with or without ulceration, respectively. These patients have an unmet clinical management need as there is no clear evidence for effective systemic adjuvant therapy to prevent disease recurrence once the primary tumour has been completely resected, which is the current standard of care for these patients. Approximately 15% to 20% of patients diagnosed with Stage IIB and 30% of patients diagnosed with Stage IIC melanoma will have a recurrence of their melanoma at 24 months. Within 5 years of surgical resection, approximately 25% of patients with Stage IIB disease and 40% of patients with Stage IIC disease will have disease recurrence. Among patients with stage IIB and IIC melanoma local recurrence occurs in 19 and 11% respectively; 45 and 58% experience regional recurrence and 44 and 39% have distant recurrence.

Patients who present with localized disease and primary tumours of less than 2.0 mm with ulceration (T2b), or primary tumour of >2.0 to 4.0 mm without ulceration (T3a) are categorised as having stage IIA melanoma. A subset of these patients have a high risk of recurrence and may benefit from adjuvant treatment. Melanoma Institute Australia has developed a risk prediction tool which will be used to select this additional high-risk population (i.e., those predicted to be at ≥ 20% recurrence at 5 years, melanomarisk.org.au). The high-risk group is identified using the following variables: mitotic rate, (count) presence of ulceration (yes/no), Breslow thickness (mm), lymphovascular invasion (present vs. absent), SNB status (negative vs not known), presence of tumour infiltrating lymphocytes (TILs), age (years), and sex (male vs. female).

The concept of moving immunotherapies from a more advanced setting where their efficacy has been well established, into a setting of stage II disease is well supported by the documented safety and efficacy data of these agents in the adjuvant setting. Introducing systemic treatment earlier in stage II disease is key to improving long term outcomes, but risk stratification is needed to identify those at most risk and manage the risk/benefit ratio given the potential immune-related toxicities.

Neoadjuvant therapy (NAT) in melanoma (and several other solid tumours) is an area of active investigation with numerous completed and ongoing trials studying a variety of therapeutic interventions utilizing diverse designs. Neoadjuvant immunotherapy and targeted therapies results in a high recurrence-free survival rate (2-year RFS >95%) for pathological responders in stage III melanoma. Subsequent management can be personalised based on the neoadjuvant response to therapy and safely provides large amounts of tissue for analysis of resistance mechanisms from those who do not have a pathological response. The neoadjuvant platform also allows for the rapid testing of novel drug combinations informing decisions to proceed to phase III trials.

Given the similar outcomes with stage III melanoma, the findings from Keynote-716, and the positive results from neoadjuvant immunotherapy trials in stage III disease, introducing neoadjuvant therapy for stage IIB/C melanoma is an opportunity to improve outcomes with 2 doses of treatment 4 weeks apart. The pathological response to immunotherapy may aid the risk stratification and identification of which patients may benefit from adjuvant therapy. The pathological response to treatment is measured by the amount of residual, viable tumour tissue in the resected specimen. In accordance with the International Neoadjuvant Melanoma Consortium criteria, a complete pathological response (pCR) is demonstrated by the complete absence of residual viable tumour cells; a near pCR is <10% of residual tumour; a partial pathological response (pPR) is 10%-50% residual tumour and no pathological response (pNR) is the presence of >50% tumour cells.

Dual checkpoint inhibition with the distinct checkpoint inhibitors relatlimab and nivolumab results in enhanced T-cell effector function that is greater than the effects of either antibody alone in murine syngeneic tumour models. The ability of anti-LAG-3 to synergize with anti-PD-1 supports the utility of combined LAG-3 and PD-1 blockade. Anti-PD-1 has already demonstrated potent anti-tumour activity in multiple human malignancies, and it is envisaged that LAG-3, when co-administered with anti-PD-1, will enhance the anti-tumour responses and potentially broaden the spectrum of tumours responsive to anti-PD-1 treatment with an acceptable safety profile.

High risk stage IIA and stage IIB/C resected melanoma represents a population of high unmet need due to the potential for locoregional, nodal or systemic recurrence, which dramatically impacts post-recurrence survival, especially in the case of systemic recurrences. Patients with stage IIB/IIC disease have a thick or ulcerated primary melanoma, with a 10-year overall survival (OS) of 82% and 75%, respectively, similar to that seen in stage IIIA and IIIB melanoma (88% and 77% respectively). In Australia, the current recommended standard of care for patients diagnosed with AJCC (8th edition) Stage IIB/C melanoma is observation.

The robust clinical activity demonstrated by nivolumab and relatlimab in patients with stage III and advanced melanoma, the manageable safety profile, and the lack of standard of care for patients who are at high risk for recurrence after a complete surgical resection of select stage IIA and stage IIB/IIC melanoma supports the further development of this drug combination in this population of patients.

Based upon the improvements seen in PFS with the addition of relatlimab to nivolumab in RELATIVITY 047 and major pathological responses in neoadjuvant treatment of stage III melanoma, this study will investigate the pathological response to 2 doses of this novel combination immunotherapy (on days 1 and 294) in patients with AJCC stage IIB and IIC melanoma (i.e. stage II based on biopsy of the primary melanoma and a clinically negative [CT and ultrasound scan assessed] regional lymph node basin(s)). Melanoma Institute Australia's risk prediction tool will be used to select an additional high risk population from those with AJCC stage IIA melanoma in need of adjuvant treatment (i.e., those predicted to be at ≥ 20% recurrence at 5 years (melanomarisk.org.au).

Neoadjuvant treatment will be followed by sentinel lymph node biopsy and complete surgical excision of the primary lesion at 6 weeks. Patients who have a pCR or near-pCR will undergo surveillance only. Remaining patients will receive adjuvant treatment with relatlimab 160 mg and nivolumab 480 mg every 4 weeks for 11 cycles (for an overall total of 13 cycles). Translational studies will be performed on tissue, blood and stool samples collected at baseline and at week 6 to identify potential predictors or response to drug and identification of potential biomarkers of recurrence. Data on the mechanisms of resistance to systemic therapies using tumour and liquid biopsy samples may lead to innovative treatment strategies to prevent resistance and improve outcomes in both the adjuvant and metastatic settings. Patients will be followed up for recurrence and survival for 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. The patient (or legally acceptable representative, if applicable) provides written informed consent for the trial.
2. Male/female patients who are at least 18 years of age on the day of signing informed consent.
3. Histologically confirmed primary cutaneous melanoma from a partial core biopsy, punch biopsy, or excisional biopsy with residual macroscopic disease.
4. AJCC (8th edition) clinical stage IIB (T3b and T4a) or IIC (T4b) melanoma, or stage IIA (T2b and T3a) melanoma with a ≥ 20% risk of recurrence at 5 years according to the MIA stage II risk calculator (melanomarisk.org.au).
5. Synchronous primaries are acceptable if there is certainty that a lesion does not represent in-transit disease and consideration should be given to the need for multiple lymph mapping requirements.
6. Past history of a primary melanoma that has been completely excised. If a patient had an SNB, this must be negative.
7. Locoregional, nodal or metastatic spread must be ruled out with clinical examination, dermoscopy, RCM and LC-OCT, CT, MRI (or CT) brain, PET, SPECT/CT and lymphoscintigraphy (including ultrasound of draining nodal basin(s)). Patients with demonstrated clinical stage III melanoma are not eligible.
8. BRAF / NRAS mutant or wild type melanoma included.
9. Availability of the diagnostic tumour sample for translational studies.
10. Surgery has been planned for sentinel node biopsy and complete resection of stage II disease. Only cases where a complete surgical resection leading to tumour free margins and which can be safely achieved without being overly morbid is considered "resectable". Resectability of each case has been agreed upon within the context of a Multi-Disciplinary Team (MDT) meeting.
11. Eastern Cooperative Oncology Group (ECOG) status 0 to 1.
12. Adequate haematological, hepatic, renal and endocrine function on blood pathology testing.
13. Anticipated life expectancy of >12 months.
14. Agreement to avoid pregnancy for the duration of treatment: Women of childbearing potential (WOCBP) must not be breastfeeding and must have a negative pregnancy test within 3 days prior to initiation of dosing. She must agree to use an acceptable method of birth control from the time of the negative pregnancy test, through the duration of treatment with the study combination plus 5 half-lives of study treatment for a total of 5 months post-treatment completion.

Exclusion Criteria:

1. Clinical or radiographic evidence of nodal, in-transit, satellite or microsatellite metastases or distant melanoma metastases.
2. Any contraindication to the administration of relatlimab or nivolumab.
3. A history of allergy or hypersensitivity to study treatment components.
4. Prior immunotherapy for any malignancy (including, but not limited to: anti-PD-1, CTLA-4, PDL-1 or anti-LAG3 or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways).
5. Patients with a condition requiring chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of study treatment. The following are permitted:

   1. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc)
   2. Inhaled or intranasal corticosteroids (with minimal systemic absorption) may be continued if patient is on a stable dose
   3. Non-absorbed intra-articular steroid injections.
6. Has active autoimmune disease that has required systemic treatment in the past 12 months (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). The following are permitted:

   1. Vitiligo
   2. Type I diabetes mellitus
   3. Residual autoimmune hypothyroidism on stable hormone replacement
   4. Resolved childhood asthma or atopy
   5. Psoriasis not requiring systemic treatment
   6. Autoimmune conditions which are not expected to recur in the absence of an external trigger.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. The following malignancies, if undergone successful definitive resection or curative treatment, are permitted:

   1. Basal cell carcinoma of the skin
   2. Squamous cell carcinoma of the skin
   3. Carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy)
   4. Prostatic intraepithelial neoplasia
   5. Atypical melanocytic hyperplasia
   6. Other malignancies for which the patient has been disease free for 1 year.
8. Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

   1. Myocardial infarction or stroke/transient ischemic attack within the 6 months prior to consent
   2. Uncontrolled angina within the 3 months prior to consent
   3. Any history of clinically significant arrhythmias (such as poorly controlled atrial fibrillation, ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
   4. QTc prolongation > 480 msec
   5. History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, poorly controlled venous thrombosis, etc)

   (g) Cardiovascular disease-related requirement for daily supplemental oxygen (h) History of 2 or more M.I.s OR 2 or more coronary revascularization procedures (regardless of the number of stent placements during each procedure) (i) Patients with history of myocarditis, regardless of aetiology.
9. Troponin T (TnT) or I (TnI) >2 × institutional ULN. Participants with TnT or TnI levels between >1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤1 ULN. If TnT or TnI levels are between >1 to 2 × ULN within 24 hours, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are <2 × ULN, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. Notification of the decision to enrol the participant following cardiologist recommendation has to be made to the Investigator,
10. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis or current interstitial lung disease.
11. Has an active infection requiring systemic therapy.
12. Treatment with complementary medications (e.g., herbal supplements or traditional Chinese medicines).
13. Any live / live-attenuated vaccine (e.g., varicella, zoster, yellow fever, rotavirus, oral polio and measles, mumps, rubella [MMR]) within 30 days of first study treatment, during treatment and until 135 days post last dose. Inactivated / killed vaccines are permitted..
14. Active SARS-CoV-2 infection. The following are permitted

    1. At least 10 days (4 weeks for severe/critical illness) have passed since symptoms first appeared or positive RT-PCR or viral antigen test result.
    2. At least 24 hours have passed since the last fever without the use of fever-reducing medications.
    3. Acute symptoms (e.g., cough, shortness of breath) have resolved.
    4. In the opinion of the investigator, there are no COVID-19-related sequelae that may place the participant at a higher risk of receiving study treatment.
    5. Recommended negative follow-up SARS-CoV-2 RT-PCR or viral antigen test based on institutional / local guidelines.
15. Has a known history of Human Immunodeficiency Virus (HIV). Note: no testing for HIV is required unless mandated by local health authority.
16. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
17. Has a known history of active TB (Bacillus Tuberculosis).
18. Pregnant or breast feeding females.
19. Concurrent medical or social conditions that may prevent the patient from attending assessments per schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2035-10 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | Week 6
  The primary endpoint is the pathological response rate at surgery (between days 43 and 56) from the first dose of neoadjuvant study treatment. The pathological response is categorised thus:
  * Complete pathological response (pCR) - 0% viable tumour cells in the surgical specimen
  * Near complete pathological response - (near pCR) - <10% viable tumour
  * Partial pathological response (pPR) - 10%-50% viable tumour
  * No pathological response (pNR) - >50% viable tumour
  The proportion of participants with a pCR, or near pCR will determine the pathological response rate.
Feasibility of recruitment | 2 years
  1. Proportion of patients enrolled in the study from the population of patients presenting to the clinic with new stage II disease, and the reason(s) for exclusion.
  2. The proportion of stage II patients with residual disease following diagnostic biopsy.
  3. Proportion of eligible patients who consent to the study.
  4. The number of patients recruited per month compared to the expected 20 patients over 24 months or 0.84 per month.

SECONDARY OUTCOMES:
The positive sentinel node biopsy rate at surgery at week 6 | Week 6
  1. The proportion of patients undergoing a sentinel node biopsy who have a positive result in the lymph node.
  2. The number of sentinel nodes identified and the number harvested.
  3. The proportion of patients with a positive sentinel node biopsy who undergo complete lymph node dissection.
The difference in sentinel lymph node (SLN) mapping between baseline and surgery at week 6. | Week 6
  The proportion of patients with the earliest EFS outcome of:
  1. The number and location of SLN identified at both timepoints.
  2. The number of baseline SLN not present at week 6.
  3. The number of new SLN at week 6.
  4. Concordance rate of SLN mapping pre- versus post-neoadjuvant therapy.
  5. Positivity rate in SLN pre- versus post-neoadjuvant therapy.
The melanoma-related event-free survival (EFS). | 10 years
  The proportion of patients with the earliest EFS outcome of any of the following events:
  1. Melanoma progression, from the initiation of study treatment prior to planned surgery (leading to unresectable stage III or stage IV disease).
  2. Melanoma recurrence, from the date of surgery (local, regional or distant).
  3. Study treatment-related death from the initiation of study treatment.
  4. Melanoma-related death, from the initiation of study treatment.
Recurrence-free survival | From surgery to 10 years
  The proportion of patients with an histologically confirmed diagnosis of disease recurrence (local, regional, and distant), as detected by the patient, on physical examination or during imaging surveillance, or death from any cause.
Overall survival | 10 years
  The proportion of participants deceased from any cause.
Safety and tolerability of neoadjuvant and adjuvant treatment and surgical procedures. | 100 days from last dose of study treatment
  The proportion of patients with adverse events as described in CTCAE version 5.0
To assess surgical outcomes following neoadjuvant therapy | Baseline and Week 6
  A comparison of expected surgical outcomes at baseline to those reported at week 6 per modified International Neoadjuvant Melanoma Consortium questionnaires.
Recurrence of melanoma in the lymph node basin where the sentinel lymph node was biospied at week 6 | 1 year from surgery
  The incidence of a recurrence of melanoma in the lymph node basin where the sentinel lymph node was mapped at baseline and biopsied at week 6.
Patient reported quality of life | 1 year
  The individual, summary and composite scores obtained from the validated EUROQOL QLQ-C30, EQ-5D, FACT-M and MCQ-28 questionnaires.
Biomarker analyses | 10 years
  Identification of predictive or prognostic biomarkers from tumour and blood analyses at baseline, surgery and at recurrence, and correlated with pathological and clinical response and toxicity.
Microbiome analyses | 10 years
  From serial faecal samples and a baseline urine sample (testing gut permeability)
  1. Correlation of bacterial diversity and abundance with treatment response and incidence of treatment-related toxicities.
  2. Correlation of self-reported dietary habits (including use of oral probiotics) at baseline and impact on bacterial diversity in the gut.
  3. The use of antibiotics during neoadjuvant treatment and the impact on intestinal bacterial diversity and abundance.
  4. Correlation of gastrointestinal mucosal integrity with bacterial composition in stool samples and immune related adverse events and response.
Change in dermoscopy, reflectance confocal microscopy (RCM) and line field confocal optical coherence tomography (LC-OCT) images during neoadjuvant treatment. | Week 6
  1. Changes from baseline dermoscopy and photography to week 4 and to week 6 including: size of lesion(s), change in colour, morphological changes.
  2. Changes from baseline RCM and LC-OCT to week 6 including: microscopy cellular resolution, tumour infiltrating lymphocytes, neovascularisation, pigment laden macrophages margin.
  3. Difference between dermoscopy, RCM and LC-OCT at each timepoint (as above).
  4. Correlation of dermoscopy, RCM and LC-OCT with histopathology findings at baseline and week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Georgina Long, Principal Investigator — Melanoma Institute Australia
Locations (1):
- Melanoma Institute Australia, Wollstonecraft, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided